CLINICAL TRIAL: NCT00514358
Title: A Multicenter, Open Label Pharmacokinetic Study of Fluconazole in Infants
Brief Title: Fluconazole Pharmacokinetics in Infants
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Pediatric Pharmacology Research Units Network (Network)
Responsible Party: Kelly Wade, MD PhD, Children's Hospital of Philadelphia
Other Study IDs: PPRU10826
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Fungal Infection
Keywords: Fungal; Infection; sepsis; pharmacokinetics
MeSH Terms: conditions — Mycoses; Infections; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- gestational age

SUMMARY:
The purpose of this study is to determine the pharmacokinetics of fluconazole in infants and evaluate the dose exposure relationship of current fluconazole dosing in infants who are receiving fluconazole for the prevention or treatment of systemic fungal infections.

DETAILED DESCRIPTION:
Systemic fungal infections in neonates are associated with high morbidity and mortality. The increasing use of intravenous central catheters, parenteral nutrition, and antibiotics in neonatal intensive care units has contributed not only to improved survival but also to the increasing incidence of fungal sepsis particularly in preterm infants. Decreasing fungal colonization can decrease the risk of systemic fungal infection. Fluconazole is a potent antifungal agent in the triazole family. Fluconazole has been shown to reduce the risk of fungal colonization and systemic infection however we do not have sufficient pharmacokinetic information in neonates to support dosing guidelines. In this study, we will perform a population pharmacokinetic study in neonates receiving fluconazole as standard of care. Fluconazole levels will be measured using a liquid chromatography/tandem mass spectroscopy (LC/MS/MS) assay from very small quantities of blood appropriate for neonates. Pharmacokinetic data obtained in this study will support appropriate dosing of fluconazole in neonates and provide information regarding drug metabolism in neonates.

ELIGIBILITY:
Inclusion Criteria:

1. Infant born >23 weeks gestational age with postnatal age <120 days
2. Due to receive fluconazole therapy for clinical care
3. Permission from attending neonatologist
4. Informed consent of parent or legal guardian

Max Age: 119 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature and term infants less than 90 days of age who are receiving fluconazole as standard of care therapy.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To develop a population PK model of fluconazole drug disposition in premature infants who are receiving fluconazole for treatment or prophylaxis against systemic fungal infections. | 3 weeks
  PK blood samples obtained over 3 weeks in infants receiving fluconazole as standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Kelly C. Wade, M.D., Ph.D., Principal Investigator — Children's Hospital of Philadelphia; Peter C Adamson, M.D., Principal Investigator — Children's Hospital of Philadelphia; Jeffery Barrett, Ph.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (5):
- United States (5):
  - Children's Hospital of Michigan, Wayne State University, Detroit, Michigan
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Result] Wade KC, Benjamin DK Jr, Kaufman DA, Ward RM, Smith PB, Jayaraman B, Adamson PC, Gastonguay MR, Barrett JS. Fluconazole dosing for the prevention or treatment of invasive candidiasis in young infants. Pediatr Infect Dis J. 2009 Aug;28(8):717-23. doi: 10.1097/INF.0b013e31819f1f50. PMID 19593252
- [Result] Wade KC, Wu D, Kaufman DA, Ward RM, Benjamin DK Jr, Sullivan JE, Ramey N, Jayaraman B, Hoppu K, Adamson PC, Gastonguay MR, Barrett JS; National Institute of Child Health and Development Pediatric Pharmacology Research Unit Network. Population pharmacokinetics of fluconazole in young infants. Antimicrob Agents Chemother. 2008 Nov;52(11):4043-9. doi: 10.1128/AAC.00569-08. Epub 2008 Sep 22. PMID 18809946